CLINICAL TRIAL: NCT04906031
Title: Sodium Stibogluconate in the Myelodysplastic Syndromes/Acute Myeloid Leukemia With One of the 65 Defined p53 Mutations That Can be Functionally Rescued by Sodium Stibogluconate
Brief Title: Sodium Stibogluconate in the MDS/AML With One of the 65 Defined p53 Mutations
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital of Jinan University (Other)
Collaborators: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Hui Zeng, Director of Hematology Department of the First Affiliated Hospital of Jinan University, First Affiliated Hospital of Jinan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FirstJinanU_SSG
Record Dates: First submitted 2021-05-18; First posted 2021-05-28 (Actual); Last update posted 2021-06-09 (Actual); Status verified 2021-06

CONDITIONS: Myelodysplastic Syndromes; Acute Myeloid Leukemia; Myeloid Malignancy; Temperature-Sensitive p53 Mutation; Sodium Stibogluconate; P53 Mutation
Keywords: Myelodysplastic Syndromes; Acute Myeloid Leukemia; Myeloid Malignancy; Temperature-sensitive p53 Mutations; Sodium Stibogluconate; p53; precision medicine; antimonial
MeSH Terms: conditions — Myelodysplastic Syndromes; Leukemia, Myeloid, Acute | interventions — Antimony Sodium Gluconate

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sodium stibogluconate (Experimental): Sodium stibogluconate 900 mg/m2/day will be given on d1-5 and d15-19. 28 days per cycle.
  Interventions: Drug: Sodium stibogluconate

INTERVENTIONS:
Drug: Sodium stibogluconate — Sodium stibogluconate 900 mg/m2/day will be given on d1-5 and d15-19. 28 days per cycle.
  Other Names: SSG

SUMMARY:
To evaluate the safety and effectiveness of Sodium Stibogluconate in the treatment of myelodysplastic syndrome/acute myeloid leukemia (MDS/AML) with p53 mutation from a defined list. The list includes 65 p53 mutations that were experimentally confirmed to be pharmacologically restored with tumor-suppressive function by antimonials.

DETAILED DESCRIPTION:
p53 is inactivated by over hundreds of diverse mutations in cancer. The investigator purposefully selected the phenotype-reversible temperature-sensitive (TS) p53 mutations for pharmacological rescue, and pertinently used p53 thermostability as readout to screen for TS p53 mutation rescue compounds. By this, the investigator identified antiparasitic drug antimonials efficiently thermostabilized the TS mutants by noncovalent binding. The antimonials met the three go-to criteria as a targeted drug-availability of co-crystal structure, structure model-compatible Structure-Activity Relationship, and target (p53)-specificity in cells, and consequently extended survival of xenograft mouse with TS p53 mutant.

Under the clinical antiparasitic dosage, the antimonials effectively rescued TS p53 mutant in patient-derived primary acute myeloid leukemia cells. Scan of the most frequent 815 p53 missense mutations identified 65 of them, predominantly TS mutations, as the antimonial-treatable mutations. Thus, the trial aims to evaluate the safety and effectiveness of the approved antimonial-Sodium Stibogluconate-in the treatment of myelodysplastic syndrome/acute myeloid leukemia (MDS/AML) with the 65 antimonial-treatable p53 mutants.

ELIGIBILITY:
Inclusion Criteria:

1. Pathologically confirmed myelodysplastic syndrome (MDS) or acute myeloid leukemia (AML).
2. Patients with one of the 65 antimonial-treatable p53 mutations with > 5% VAF: Q136P, Y234H, V272M, F270V, P278A, R213L, Y126H, T253N, T253I, R158L, Q136E, P142F, A129D, L194R, R110P, V172G, C176F, I254N, K305R, E285D, T155P, H296D, E258G, G279V, T211A, R213P, C229Y, I232F, E294K, P152R, R196P, M160T, N131S, N131H, K139N, L330H, Y220N, E298Q, D148E, L264R, E224D, H168P, N263H, K320N, S227C, E286D, K292T, V203A, M237R, F212L, K132Q, Y236S, Y126S, Q136H, E221A, I232S, Y163H, P190T, C182Y, P142L, Y163S, V218E, I195S, V272A, and S106R.
3. Life expectancy >12 weeks.
4. ECOG Performance status < 3.
5. Aged from 18 to 75.
6. Active bone marrow hyperplasia indicated by morphology.
7. Normal liver and renal function, bilirubin ≤35μmol/L, ASL/ALT lower than 2xULN, creatinine level ≤150μmol/L.
8. Normal cardiac function.
9. Lung function: dyspnea ≤ CTC AE grade 1 and SaO2≥ 92% in indoor air environment.
10. Written Informed consent.

Exclusion Criteria:

1. Confirmed CNS involvement.
2. Severe cardiac diseases including myocardial infarction or heart insufficiency.
3. QT interval ≥450ms on ECG.
4. With other visceral malignancy.
5. Active tuberculosis or HIV(+).
6. Patients with pregnancy or lactation.
7. Allergic or significantly contraindicated to any drugs involved in intervention.
8. Previous intolerance or allergy history to similar drugs.
9. Participation at same time in another study in which investigational drugs are used.
10. Any other conditions interfering the study.
11. Abnormal liver function which does not meet the inclusion criteria.
12. ECOG performance status ≥3, CCI >1, ADL <100.
13. Aged <18 years or >75years

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2023-02-01 (Estimated); Study Completion 2024-02-01 (Estimated)

PRIMARY OUTCOMES:
Overall response rate | At the end of Cycle 4 (each cycle is 28 days)
  Partial response (PR) + complete response (CR) rate

SECONDARY OUTCOMES:
Adverse Event (AE) | At the end of Cycle 4 (each cycle is 28 days)
  Adverse events (AEs) will be reported and graded

CONTACTS AND LOCATIONS:
Overall Officials: Min Lu, PHD, Principal Investigator — Ruijin Hospital
Locations (1):
- First Affiliated Hospital of Jinan University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Tang Y, Song H, Wang Z, Xiao S, Xiang X, Zhan H, Wu L, Wu J, Xing Y, Tan Y, Liang Y, Yan N, Li Y, Li J, Wu J, Zheng D, Jia Y, Chen Z, Li Y, Zhang Q, Zhang J, Zeng H, Tao W, Liu F, Wu Y, Lu M. Repurposing antiparasitic antimonials to noncovalently rescue temperature-sensitive p53 mutations. Cell Rep. 2022 Apr 12;39(2):110622. doi: 10.1016/j.celrep.2022.110622. PMID 35417717